CLINICAL TRIAL: NCT04913454
Title: CLearing Alzheimer's Disease Molecular Pathology Without Medications
Acronym: CLAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Daniele Altomare, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00989
Record Dates: First submitted 2021-05-25; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease; Amyloid Plaque; Amyloidosis
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Amyloidosis | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training (Experimental): 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training (1 hour/day, per 5 days/week, for a total of 8 weeks).
  Interventions: Other: 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training
- Cognitive training only (Active Comparator): Cognitive training only (1 hour per day, per 5 days/week, for a total of 8 weeks).
  Interventions: Other: Cognitive training

INTERVENTIONS:
Other: 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training — 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training (1 hour/day, per 5 days/week, for a total of 8 weeks)
  Arms: 40 Hz multi-sensory (auditory + visual) stimulation and cognitive training
Other: Cognitive training — Cognitive training (1 hour/day, per 5 days/week, for a total of 8 weeks)
  Arms: Cognitive training only

SUMMARY:
According to the most popular pathophysiological models of Alzheimer's disease, the amyloid hypothesis, amyloid deposition is the causative event triggering a chain of other downstream events which finally lead to Alzheimer's disease and dementia. In mouse models of Alzheimer's disease, 40 Hz multi-sensory (auditory and visual) stimulation was able to reduce the number and size of amyloid plaques throughout cortex and improve cognitive performance.

The primary objective of this study is to assess whether an intervention consisting of 40 Hz multi-sensory (auditory and visual) stimulation is able to reduce the amyloid load in non-demented amyloid-positive individuals.

As secondary objectives, the investigators will assess whether such intervention is able to:

* improve the brain electrical activity,
* improve or slow down the worsening of Alzheimer's blood-based biomarkers,
* improve or slow down the worsening of cognition.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form),
* age 40-80,
* ≥5 years of education,
* previous evidence of brain amyloidosis (assessed by PET, CSF, or blood-based biomarkers).

Exclusion Criteria:

* history of epilepsy;
* clinically relevant visual or auditory diseases/deficits;
* clinical diagnosis of dementia;
* contraindication to amyloid-PET;
* inability to undergo the procedures of the study, e.g. severe behavioral disturbances;
* severe diseases:

  1. Malignant neoplasm within 5 years,
  2. Life threatening diseases,
  3. Severe systemic diseases (e.g. kidney insufficiency, cardiac insufficiency, decompensated diabetes, decompensated metabolic diseases, decompensated hypothyroidism, uncontrolled autoimmune diseases);
* the participation to a clinical trial involving potential Alzheimer's disease modifying therapies;
* documented pregnancy or intention to become pregnant during the course of the study or breast feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in amyloid load | 8 weeks
  Changes in amyloid load assessed by longitudinal amyloid-PET

SECONDARY OUTCOMES:
Changes in brain electrical activity | 8 weeks
  Changes in brain electrical activity (e.g. gamma power spectral density) assessed by longitudinal EEG
Changes in Alzheimer's blood-based biomarkers | 8 weeks
  Changes in Alzheimer's blood-based biomarkers (e.g. plasma Aβ42/Aβ40 ratio, Aβ42, Aβ40, p-tau, and neurofilament light) assessed by longitudinal blood sample collection
Changes in cognition | 8 weeks
  Changes in cognition (using the Preclinical Alzheimer Cognitive Composite (PACC) score) assessed by longitudinal neuropsychological assessment

IPD SHARING:
Plan to Share IPD: Undecided